CLINICAL TRIAL: NCT04716491
Title: Promotion of Sleep for Patients Submitted to Percutaneous Intervention to Treat Heart Diseases: Randomized Clinical Trial
Brief Title: Promotion of Sleep for Patients Submitted to Percutaneous Intervention to Treat Heart Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Regina Claudia da Silva Souza, Master, Hospital Sirio-Libanes
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: AVAP-NG 1527
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Sleep Hygiene
Keywords: Sleep Deprivation; Intensive Care Units
MeSH Terms: conditions — Sleep Hygiene; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: The sample will be divided into two groups: intervention group (formed by participants who will wear eye masks and hearing protectors) and control group (formed by participants who will not use any device, that is, they will receive the usual care of the unit that does not include any sleep hygiene approach)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The main researcher will not participate in the recruitment, application of the intervention and data collection steps. There will be interventional nurses who have been trained by them and who will do these actions.The outcomes defined at the beginning of the study will be analyzed by a statistician who will not participate in the randomization process and in any step prior to data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention to decrease disruptive sleep in patients undergoing percutaneous intervention to treat cardiac disorders admitted to the ICU: ear protector and eye mask.
  Interventions: Device: Intervention to decrease disruptive sleep in patients undergoing percutaneous intervention to treat cardiac disorders admitted to the ICU: ear protector and eye mask.
- Control group (No Intervention): Participants will not use the devices at any time of admission to the intensive care unit

INTERVENTIONS:
Device: Intervention to decrease disruptive sleep in patients undergoing percutaneous intervention to treat cardiac disorders admitted to the ICU: ear protector and eye mask. — When they meet the inclusion criteria and accept to participate in the study, the interventionist nurse will explain to the patient the objectives and protocol of the study, apply the consent form and the instruments for assessing sleep (pittsburgh), trait and state anxiety (STAI). Then the software will be randomized and after defining the group, the nurse will guide the patient on the use of the devices from 9:00 am until the final awakening in the morning. Control group participants will only complete the assessment instruments. Noise and brightness will be measured at randomization of participants. The following morning, the visual sleep scale and the sleepiness scale will be applied for both groups, in addition to filling in information regarding the length of time the devices stay with patients at night and the clinical data that will be collected until discharge from the hospital. ICU, when independent of the group, the state anxiety instrument will be applied.
  Arms: Intervention group

SUMMARY:
Patients undergoing treatment for heart disease through percutaneous interventions admitted to intensive care units often suffer from sleep deprivation, with multifactorial factors being the precursors of this problem. Sleep deprivation has a negative impact on rehabilitation, with increased morbidity and mortality. Therefore, implementing non-pharmacological measures for this population is essential for better quality care, as well as more satisfactory experiences. The Objectives are to evaluate whether the non-pharmacological intervention that includes the use of eye masks and hearing protectors has an influence on the quality of sleep of patients undergoing percutaneous interventions for the treatment of heart diseases admitted to the intensive care unit, to compare the quality of sleep between patients according to sociodemographic and clinical variables and to identify whether anxiety is a factor associated with sleep quality in patients undergoing percutaneous interventions for the treatment of heart disease in patients admitted to the intensive care unit. Randomized clinical trial blinded to the steps of data collection and data analysis, with two groups of participants in which the intervention with eye masks and ear protectors will be evaluated. The inclusion criteria in the study will be patients undergoing percutaneous intervention treatment for heart disease over the age of 18, preserved communication skills and understanding. The study site will be a cardiac intensive care unit in a private hospital of high complexity in the city of São Paulo. The intervention will be carried out during the period of hospitalization in the intensive care unit, by nurses trained by the researcher from 9 pm until the patient awakens, and variables related to sleep quality, anxiety, pain, delirium and length of stay will be collected. in bed. The sample will consist of 80 patients divided into two groups (intervention and control) and the data will be analyzed with descriptive statistics, with Student t test and Mann Whitney test for comparison between groups and with Chi-square test and Spearman for analysis of categorical variables. . Relative risk, odds ratio will be calculated and the level of significance adopted will be 5%. It is intended to know if the non-pharmacological intervention brings benefits to reduce sleep deprivation and contributes to better clinical outcomes.

DETAILED DESCRIPTION:
The intervention to promote sleep in patients undergoing percutaneous intervention to treat cardiac disorders admitted to the ICU will be the use of ear protectors and eye masks. The purpose of the intervention is to promote sleep in this population by reducing noise and light in the Intensive Care Unit environment. The devices used will be the use of black silk masks with elastic for protection of the eyes against light and a silicone ear protector to reduce environmental noise. The procedure will consist of the following steps: application of the free and informed consent form, sleep assessment instruments, trait and state anxiety and collection of sociodemographic and clinical data and randomization in the arms of the study at the patient's admission to the ICU, guidance on the use of devices from 21 hours and until awakening, measurement of noise and brightness at the time of placing the devices, application of the visual sleep scale in the morning during the physical examination, note every two hours on a specific form whether the patient remains with the devices. These steps will be performed by the interventionist nurses who will be trained by the main researcher and will approach the patients in the inpatient unit or in the Intensive Care Unit after admission.

The intervention will be applied only in the Cardiac Intensive Care Unit, and after discharge from the ICU, patients will be able to use it if they want the devices to sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Have the ability to communicate verbally and understand what is requested in the assessment instruments, according to the nurse's initial assessment performed on admission.

Exclusion Criteria:

1. Report of a serious sleep disorder that requires daily treatment before hospitalization, such as sleep apnea, narcolepsy and chronic insomnia.
2. Presence of severe complication (aortic dissection, bleeding or stroke after the procedure) related to the treatment.
3. Presence of delirium as assessed in the medical record.
4. Severe hearing and visual loss.
5. History of neurological disease or diagnosed psychiatric disorders.
6. Admission to the Intensive Care Unit between the hours of 9:00 pm to 6:00 am after the percutaneous intervention procedure.
7. Treatment with mechanical ventilation.
8. Need for sedation while in the ICU.
9. Who are not fluent in the Portuguese language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | During the patient's stay in the ICU until discharge from the unit during the patient's stay in the ICU until discharge from the unit for about three months
  Sleep quality will be assessed by the visual sleep scale, adapted and validated in Brazil from the original instrument Verran Snyder-Halpern Sleep Scale that allows daily self-assessment of the sleep efficiency of hospitalized patients regarding their last night of slep

SECONDARY OUTCOMES:
Sleepiness | During the patient's stay in the ICU until discharge from the unit during the patient's stay in the ICU until discharge from the unit for about three months
  The Epworth Excessive Sleepiness Scale (ESS) will be used in the morning to allow the patient to self-assess the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Regina Souza, master, Principal Investigator — Hospital Sirio-Libanes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beltrami FG, Nguyen XL, Pichereau C, Maury E, Fleury B, Fagondes S. Sleep in the intensive care unit. J Bras Pneumol. 2015 Nov-Dec;41(6):539-46. doi: 10.1590/S1806-37562015000000056. PMID 26785964
- [Background] Cicek HS, Armutcu B, Dizer B,Yava A, Tosun N, Celik T. Sleep quality of patients hospitalized in the coronary intensive care unit and the affecting factors. International Journal of Caring Sciences. 2014;7(1):324-32.
- [Background] Machado FS, Souza RCDS, Poveda VB, Costa ALS. Non-pharmacological interventions to promote the sleep of patients after cardiac surgery: a systematic review. Rev Lat Am Enfermagem. 2017 Sep 12;25:e2926. doi: 10.1590/1518-8345.1917.2926. PMID 28902932
- [Background] Vieira JV, Ferreira RF, Goes MP. Ear and eye protectors in the promotion of sleep in intensive care. J Nurs UFPE 2018;12(10):2784-93. https://doi.org/10.5205/1981-8963-v12i10a236958p2784-2793-2018.
- [Background] Dhooria S, Sehgal IS, Agrawal AK, Agarwal R, Aggarwal AN, Behera D. Sleep after critical illness: Study of survivors of acute respiratory distress syndrome and systematic review of literature. Indian J Crit Care Med. 2016 Jun;20(6):323-31. doi: 10.4103/0972-5229.183908. PMID 27390455
- [Background] Elliott R, McKinley S, Cistulli P. The quality and duration of sleep in the intensive care setting: an integrative review. Int J Nurs Stud. 2011 Mar;48(3):384-400. doi: 10.1016/j.ijnurstu.2010.11.006. Epub 2010 Dec 24. PMID 21185560
- [Background] Menger J, Urbanek B, Skhirtladze-Dworschak K, Wolf V, Fischer A, Rinosl H, Dworschak M. Earplugs during the first night after cardiothoracic surgery may improve a fast-track protocol. Minerva Anestesiol. 2018 Jan;84(1):49-57. doi: 10.23736/S0375-9393.17.11758-X. Epub 2017 Jul 20. PMID 28726359
- [Background] Locihova H, Axmann K, Padysakova H, Fejfar J. Effect of the use of earplugs and eye mask on the quality of sleep in intensive care patients: a systematic review. J Sleep Res. 2018 Jun;27(3):e12607. doi: 10.1111/jsr.12607. Epub 2017 Sep 25. PMID 28944590
- [Background] Sadeh A. Iii. Sleep assessment methods. Monogr Soc Res Child Dev. 2015 Mar;80(1):33-48. doi: 10.1111/mono.12143. PMID 25704734